CLINICAL TRIAL: NCT01712321
Title: Vilazodone in the Treatment of Social Anxiety Disorder: A Double Blind Study
Brief Title: Study of Vilazodone to Treat Social Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Medical Research Network (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VII-IT-07
Record Dates: First submitted 2012-10-18; First posted 2012-10-23 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Social Anxiety; Social Phobia; SAD
MeSH Terms: conditions — Phobia, Social | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vilazodone (Experimental): Vilazodone 20mg or 40mg taken once daily by mouth for up to 12 weeks
  Interventions: Drug: Vilazodone
- Placebo (Placebo Comparator): Placebo to match Vilazodone 20mg or 40mg, taken once daily by mouth for up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vilazodone — Vilazodone 20mg or 40mg taken once daily by mouth
  Other Names: Viibryd
  Arms: Vilazodone
Drug: Placebo — Placebo matching Vilazodone 20mg or 40mg, taken once daily by mouth
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Vilazodone is effective in the treatment of symptoms of Social Anxiety Disorder among adults.

DETAILED DESCRIPTION:
The proposed study is a 12 week double-blind, placebo-controlled trial in which daily doses of vilazodone 20 to 40 mg/day or matching placebo will be administered on a 1:1 ratio. The study will include 30 outpatients age 18-75 with SAD, generalized subtype who return for at least one post randomization visit where efficacy evaluations are conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Social Anxiety Disorder, generalized subtype
* LSAS total score of 70 at visits 1 and 2

Exclusion Criteria:

* Lifetime history of Bipolar disorder or Schizophrenia
* Current suicidal risk
* Current unstable medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change in Liebowitz Social Anxiety Scale (LSAS) - total score | Change from Baseline to Final Study Visit: minimum 1 week - maximum 12 weeks
  All subjects randomized to drug or placebo and returning for at least one subsequent visit will be included in the primary efficacy analyses.

SECONDARY OUTCOMES:
Responder rate, as defined by Clinical Global Impression of Improvement score of 1 or 2 | Study Endpoint: minimum 6 weeks - maximum 12 weeks
  Responder rate as defined by a CGI Improvement score of 1 (Very Much Improved) or 2 (Much Improved) at study endpoint.
  Randomized subjects taking minimum target dose (20mg or matching placebo daily) for at least six consecutive weeks will be considered a minimum adequate trial for the purposes of secondary analyses.
Change in the Clinical Global Impression of Severity of Illness score | Change from Baseline to Study Endpoint: minimum 6 weeks - maximum 12 weeks
  Randomized subjects taking minimum target dose (20mg or matching placebo daily) for at least six consecutive weeks will be considered a minimum adequate trial for the purposes of secondary analyses.
Change on the LSAS anxiety and avoidance subscales | Change from Baseline to Study Endpoint: minimum 6 weeks - maximum 12 weeks
  Randomized subjects taking minimum target dose (20mg or matching placebo daily) for at least six consecutive weeks will be considered a minimum adequate trial for the purposes of secondary analyses.
Change in Hamilton Depression scale total | Change from Baseline to Study Endpoint: minimum 6 weeks - maximum 12 weeks
  Randomized subjects taking minimum target dose (20mg or matching placebo daily) for at least six consecutive weeks will be considered a minimum adequate trial for the purposes of secondary analyses.
Change in Hamilton Anxiety scale total | Change from Baseline to Study Endpoint: minimum 6 weeks - maximum 12 weeks
  Randomized subjects taking minimum target dose (20mg or matching placebo daily) for at least six consecutive weeks will be considered a minimum adequate trial for the purposes of secondary analyses.
Subject-assessed responder rate | Study Endpoint: minimum 6 weeks - maximum 12 weeks
  Subject-assessed responder rate, as defined by a Patient Global Impression of Change score of 1 (Very Much Improved) or 2 (Much Improved) at study endpoint.
  Randomized subjects taking minimum target dose (20mg or matching placebo daily) for at least six consecutive weeks will be considered a minimum adequate trial for the purposes of secondary analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Liebowitz, MD, Principal Investigator — The Medical Research Network, LLC
Locations (1):
- The Medical Research Network, LLC, New York, New York, United States

REFERENCES:
- [Derived] Careri JM, Draine AE, Hanover R, Liebowitz MR. A 12-Week Double-Blind, Placebo-Controlled, Flexible-Dose Trial of Vilazodone in Generalized Social Anxiety Disorder. Prim Care Companion CNS Disord. 2015 Nov 26;17(6):10.4088/PCC.15m01831. doi: 10.4088/PCC.15m01831. eCollection 2015. PMID 27057414